CLINICAL TRIAL: NCT02314468
Title: Comparative Study of Negative Pressure Wound Therapy and Allogeneic Human Skin Grafts for Wound Bed Preparation in Necrotising Soft Tissue Infections
Brief Title: Negative Pressure Wound Therapy and Allogeneic Human Skin Grafts for Wound Bed Preparation
Acronym: NPWTvsGPA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/724
Record Dates: First submitted 2013-09-30; First posted 2014-12-11 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Necrotizing Soft Tissue Infection
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- negative pressure wound therapy (NPWT) (Active Comparator): negative pressure wound therapy (NPWT)
  Interventions: Procedure: Negative pressure wound therapy
- Glycerol Preserved Allografts (GPA) (Active Comparator): Glycerol Preserved Allografts (GPA)
  Interventions: Procedure: Glycerol Preserved Allografts (GPA)

INTERVENTIONS:
Procedure: Negative pressure wound therapy — NPWT changed twice a week.
  Arms: negative pressure wound therapy (NPWT)
Procedure: Glycerol Preserved Allografts (GPA) — GPA changed every 7 to 10 days.
  Arms: Glycerol Preserved Allografts (GPA)

SUMMARY:
Introduction Necrotising soft tissue infections (NSTI) incorporate a spectrum of pathologies, all characterized by an infectious state, typically arising after a penetrating trauma or a surgical procedure and an expeditious spreading of necrosis throughout the soft tissues of the body. It is a rare, life-threatening and devastating infection defined by a necrosis of fascia, subcutaneous tissues and skin. Aggressive surgical debridement to remove all necrotic tissue and define the extent of the disease is still the mainstay of correct treatment of NSTI.

Both negative pressure wound therapy (NPWT) and the application of allograft skin to debrided areas, are documented options for wound bed preparation which are standard in the university hospital of Gent.

NPWT is a technique for wound bed preparation involving the controlled application of sub-atmospheric pressure to the local wound environment, using a sealed wound dressing connected to a vacuum pump. Mechanisms of action attributed to NPWT include an increase in blood flow, promotion of angiogenesis, reduction in wound surface area, positive modulation of the inhibitory contents of wound fluid, induction of cell proliferation, reduction of edema, and bacterial clearance.

Allograft skin or cadaveric skin possesses many of the ideal properties of biologic dressings, and plays a major role in the surgical management of extensive wounds when autologous tissue may not be immediately available. It reduces evaporative water loss and the drainage of protein-rich fluids, prevents wound desiccation, and suppresses microbial proliferation. Wound pain is lessened and the allograft restores a physiologic barrier at the wound surface. Enhancing revascularization, and thereby creating a viable wound bed before final reconstruction, is perceived as one of the most important features of allografting.

DETAILED DESCRIPTION:
Study objectives This study will compare negative pressure wound therapy versus cadaveric skin as treatment options for wound bed preparation in wounds resulting from necrotising soft tissue infection.

Methodology One arm includes a NPWT system that is used in conjunction with gauze or foam dressings. Dressing changes normally will be carried out twice a week unless otherwise indicated by the wound condition, the patients clinical presentation or a seal broken beyond repair. NPWT wound bed preparation will be ended when two experienced plastic surgeons consider the wound bed suitable for autografting. (Endpoint) The second arm includes application of cadaveric skin. The allografts normally will be changed every seven to ten days or earlier depending on adhesion of the allograft to the wound bed. In practice, the ability of the allograft to adhere to the wound bed has a diagnostic value, referred to as a 'take-test'. If the allograft does not adhere, one must consider an infection or non-viable wound surface. If the allograft adheres to the wound bed and adequate granulation tissue is suspected underneath, then the wound bed is suitable for autografting. (Endpoint)

ELIGIBILITY:
Inclusion Criteria:

* Necrotising soft tissue infection

Exclusion Criteria:

None specific

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Quality of wound bed preparation until autografting. | After 3 days
  WHAT software, clinical assessment by plastic surgeon, Laser Doppler Imaging scan.

SECONDARY OUTCOMES:
Pain assessment until autografting. | After 3 days
  Numerical pain scale.
Ease of use until autografting. | After 3 days
  Numerical scale for ease of use.
Cost utility until autografting. | After 3 days
  Cost of material.

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website hospital — http://www.uzgent.be